CLINICAL TRIAL: NCT05834075
Title: A Retrospective Study to Evaluate the Early Real-world Evidence of Brolucizumab in Patients With Neovascular Age-related Macular Degeneration (nAMD) in India
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRTH258AIN02
Record Dates: First submitted 2023-04-19; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Neurovascular Age-related Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This non-interventional, retrospective, observational, noncomparative, non-randomized, single-arm, multi-centre study included patients (≥50 years) diagnosed with neovascular age-related macular degeneration (nAMD) in at least 1 eye. Anonymized data of patients treated with brolucizumab intravitreal injection (IVI) who had received the first dose of brolucizumab between 01 October 2020 and 31 March 2021 was collected. Patients could either be treatment-naïve or previously treated with single or a combination of other IVI of anti-vascular endothelial growth factors (VEGFs). The primary outcome measure was the change in fluid levels (intra-retinal fluid [IRF], sub-retinal fluid [SRF], and pigment epithelial detachment [PED]) from baseline to Month 3. Secondary outcome measures included change in best-corrected visual acuity (BCVA) and central retinal thickness (CRT), number of brolucizumab injections, and safety (number of adverse events [AEs]). Descriptive statistics were tabulated for the demographic and clinical characteristics as well as outcome variables.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naïve nAMD patients or patients previously treated with a single or a combination of other intravitreal anti-VEGFs
* Patients (male or female) ≥50 years of age at the index date
* Patients with visual acuity (VA) and optical coherence tomography (OCT) assessments at baseline and at least 1 month after initiating treatment with brolucizumab
* Patients treated with IVI of brolucizumab (received the first dose of anti-VEGF injection during the index period [01 October 2020 to 31 March 2021])

Exclusion Criteria:

* Patients with dry AMD, geographic atrophy, and other retinal diseases in the study eye
* Patients who were part of any other nAMD trial/study during the study period
* Patients undergoing additional ocular treatment along with other anti-VEGF agents

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with absence or reduction of IRF at Month 3 compared to baseline | From baseline to Month 3
  Percentage of patients with either absence of intra-retinal fluid (IRF) at Month 3 or a reduction of IRF at Month 3 compared to baseline.
Percentage of patients with absence or reduction of SRF at Month 3 compared to baseline | From baseline to Month 3
  Percentage of patients with either absence of sub-retinal fluid (SRF) at Month 3 or a reduction of SRF at Month 3 compared to baseline.
Percentage of patients with absence or reduction of PED at Month 3 compared to baseline | From baseline to Month 3
  Percentage of patients with either absence of pigment epithelial detachment (PED) at Month 3 or a reduction of PED at Month 3 compared to baseline.

SECONDARY OUTCOMES:
Mean change from baseline in BCVA at Month 3 as measured by logarithm of the minimum angle of resolution (logMAR) | Baseline and Month 3
Percentage of patients with absence or reduction of IRF at Months 1 and 2 compared to baseline | Baseline, Months 1 and 2
Percentage of patients with absence or reduction of SRF at Months 1 and 2 compared to baseline | Baseline, Months 1 and 2
Percentage of patients with absence or reduction of PED at Months 1 and 2 compared to baseline | Baseline, Months 1 and 2
Mean change from baseline in CRT at Months 1, 2, and 3 as assessed by optical coherence tomography (OCT) | Baseline, Months 1, 2, and 3
Number of brolucizumab injections during Months 1, 2, and 3 of brolucizumab treatment | Months 1, 2, and 3
Number of non-injection visits during Months 1, 2, and 3 of brolucizumab treatment | Months 1, 2, and 3
Number of visits during Months 1, 2, and 3 of brolucizumab treatment | Months 1, 2, and 3
Number of patients with treatment-emergent adverse events | Baseline to Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- India (4):
  - Narayana Nethralaya, Bangalore
  - Disha Eye Hospital, Kolkata
  - Susrut Eye Foundation and Research Center, Kolkata
  - Dr. Milan's Retina Care Center, Rajkot